CLINICAL TRIAL: NCT02783677
Title: The Application of Digital Infrared Thermal Imaging in Peripheral Artery Disease
Brief Title: The Application of Digital Infrared Thermal Imaging in Peripheral Artery Disease of the Lower Extremities
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201209053RIC
Record Dates: First submitted 2016-04-11; First posted 2016-05-26 (Estimated); Last update posted 2017-02-06 (Estimated); Status verified 2017-01

CONDITIONS: Peripheral Artery Disease; Diabetes Mellitus
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus | interventions — Angioplasty, Balloon, Coronary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- DM with PAD before angioplasty: Diabetic patients diagnosed with peripheral artery disease via vascular Duplex.
- DM without PAD: Diabetic patients diagnosed without peripheral artery disease via vascular Duplex.
- Healthy volunteers: Healthy volunteers
- DM with PAD after angioplasty: Diabetic patients diagnosed with PAD underwent balloon-angioplasty
  Interventions: Procedure: Percutaneous balloon angioplasty

INTERVENTIONS:
Procedure: Percutaneous balloon angioplasty
  Groups: DM with PAD after angioplasty

SUMMARY:
Peripheral artery disease (PAD) is highly prevalent. It occurs most often in the lower extremities. Symptoms include intermittent claudication, ischemic pain, ulceration and necrosis. Amputation may be necessary in severe cases. PAD is also an indicator of future cerebrovascular and cardiovascular events. Diabetes mellitus (DM) is one of the major risk factors of PAD. Approximately 5% to 10% of diabetic patients have had foot ulceration, and 1% have undergone amputation. Other risk factors include smoking, old age, male gender, hypertension, dyslipidemia, hyperhomocysteinemia and renal insufficiency. Ankle-brachial index (ABI) is the most popular tool used to screen PAD. Doppler-derived ankle and brachial systolic pressure is obtained. If the ratio is abnormal, further confirmation studies will necessary. Although ABI is recommended as one of the screening tests for diabetic complications in guidelines, its utility is limited in calcified non-compressible vessels, which are common in DM and renal failure patients.

Digital infrared thermal imaging (DITI) is used to detect surface temperature because objects of absolute temperatures higher than zero would radiate electromagnetic waves of certain wave lengths according to Plank's law. DITI examination is non-invasive, non-contact and fast. Theoretically, temperature of the perfusion area of the occlusive arteries will decrease. Investigators will analyze DITI of PAD, and observe the relationship between DITI, ABI and vascular duplex examination. The dynamic change of DITI before and after percutaneous transluminal angioplasty of PAD will also be observed. Investigators would like to evaluate the possibility of the clinical application of DITI for PAD screening.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20~85 years old
* Diagnosed with DM

Exclusion Criteria:

* History of lower extremities disease or underwent leg surgery
* Pregnancy
* Fever
* Leg edema
* Autoimmune disease

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with DM
Sampling Method: Non-Probability Sample
Enrollment: 230 (Estimated)
Dates: Start 2013-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Digital infrared thermal imaging (DITI) | 7 days
  Digital infrared thermal imaging (DITI) to detect surface temperature

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No